CLINICAL TRIAL: NCT05353868
Title: Gut Microbiota in the Progression of Alpha-synucleinopathies: a Prospective Follow-up Study
Brief Title: Gut Microbiota in the Progression of Alpha-synucleinopathies
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Wing Yun Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: NTEC-2021-0614
Record Dates: First submitted 2022-01-13; First posted 2022-04-29 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: REM Sleep Behavior Disorder
Keywords: Gut microbiota; Parkinson's disease; REM sleep behavior disorder
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early PD: 1. Recruited in the baseline study as a subject of the Early PD group
  2. Completed baseline assessment and stool sample collection
  3. Being capable of giving informed consent for participation of the study
  Interventions: Other: No intervention
- iRBD: 1. Recruited in the baseline study as a subject of the iRBD group
  2. Completed baseline assessment and stool sample collection
  3. Being capable of giving informed consent for participation of the study
  Interventions: Other: No intervention
- First degree relatives of patient with iRBD: 1. Recruited in the baseline study as a subject of the 'First degree relatives of patients with iRBD' group
  2. Completed baseline assessment and stool sample collection
  3. Not cohabiting with iRBD proband
  Interventions: Other: No intervention
- Health control: 1. Recruited in the baseline study as a subject of the 'healthy controls' group
  2. Completed baseline assessment and stool sample collection
  3. Being capable of giving informed consent for participation of the study
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study is to correlate baseline gut microbiota features and the progression of neurodegeneration in the established cohort of patients with early Parkinson's disease.

DETAILED DESCRIPTION:
Alpha-synucleinopathy is a major group of neurodegenerative diseases that include Parkinson's disease and Dementia of Lewy bodies. They are known to have a long preclinical development, and prodromal markers that indicate the onset of early phase of the neurodegenerative process present along the way. Among the markers, idiopathic REM sleep behavior disorder (iRBD), a distinct form of parasomnia characterised by the presence of dream-enactment behaviour and REM sleep without atonia, represent a particularly high conversion likelihood that makes it a de facto precursor of clinical diseases (14 years conversion rate >95%). Thus, RBD serves as an exclusive opportunity for us to study the early-stage progression of α-synucleinpathies, and a window for early neuroprotective intervention.

In the context of α-synucleinopathic neurodegenerative diseases, high prevalence of gastrointestinal dysfunction and the presence of alpha-synuclein aggregates in the enteric nervous system at the early stage of disease have been found. These early findings were embedded in an influential Braak's hypothesis that the process of neurodegeneration can be started by 'unknown pathogen' from gut and spread to the central nervous system via vagus nerve in a caudal-rostral manner (medulla->pon->mid/forebrain->cortex). Human data showed that microbiome composition in patient with Parkinson's disease is different from control. The relative abundance of certain microbiotas, such as Enterobacteriaceae, have been shown to be associated with the severity of motor symptoms in patients with Parkinson's disease. It is hypothesized that microbiota dysbiosis resulting in a pro-inflammatory gut environment, which in turn create excessive oxidative stress and trigger alpha-synuclein misfolding cascade. While available evidence suggests that gut-brain hypothesis potentially plays a role in the disease process of α-synucleinopathies, the exact detail of microbiota involvement will need further examination. The key question of whether microbiota dysbiosis is driving or being driven by the process of neurodegeneration, need to be answered by prospective empirical studies that examine the longitudinal course of neurodegeneration from early to late stage, and to relate such course with the corresponding dynamic profile of the subjects' gut microbiota composition. Most of the available studies on this subject were cross-sectional studies that based on patients with Parkinson's disease, the terminal stage of the neurodegenerative process. There has been only two studies that include RBD patients, suggesting some alteration of microbiota happens in RBD stage already, but the number of RBD subjects included was small (n = 21 and 26), and there was no follow-up data (10, 11). In other words, there is no study that can answer such question at the moment. This remarkable gap in literature probably reflects two major obstacles researchers would face in planning such study: the difficulties in identifying and recruiting subjects with early-stage α-synucleinopathies, and the need for sufficient follow-up period to unfold the neurodegeneration process. In this regard, the investigators investigated gut microbiota composition in our established cohort of RBD and RBD family. Preliminary finding indicated gut dysbiosis has already occurred at or likely before the onset of RBD, at an even earlier stage of synucleinopathy (i.e., high-risk relatives of RBD). For example, consistent overabundance of Ruminococcaceae UCG-002 were found in RBD relatives, patient with RBD and early PD, as compared with controls.

In this study, the investigators will perform 3-year follow-up of clinical assessments and gut microbiota measurement. The investigators aim to correlate baseline gut microbiota features and the progression of neurodegeneration, e.g., emerged autonomic dysfunctions, phenoconversion, in the established cohort of patients with early Parkinson's disease, idiopathic RBD, first-degree relatives (FDRs) of patients with iRBD and healthy controls. Besides, the investigator will examine the associations between long-term gut microbiota changes and progression of neurodegenerative biomarkers and compare the long-term changes of gut microbiota between controls and different early stages of α-synucleinopathies.

ELIGIBILITY:
Inclusion Criteria:

* recruit from the subjects who completed the baseline study

Exclusion Criteria:

* The use of probiotics or antibiotics within three months prior to sample collection;
* Pre-existing gastrointestinal diseases, such as inflammatory bowel disease.
* Not capable of giving informed consent for participation of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will recruit from the subjects who completed the baseline study, which represent different stages of α-synucleinopathies, namely patients with PD (Braak's stages 3 or 4) without dementia, patients with iRBD (Braak's stage 2), first degree relatives of iRBD patients (iRBD-FDRs, Braak's stage 0 or 1), and healthy controls (Braak's stage 0).
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Composition of gut microbiota | 2 years
  Correlation of baseline gut microbiota features and the progression of α-synucleinopathy neurodegeneration.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Data will be handled and stored under Department of Psychiatry and PI will be responsible for the safekeeping.